CLINICAL TRIAL: NCT02637492
Title: Development and Validation of a Clinical Prediction Rule for Lower Limb Critical Limb Ischaemia (PREDICCMI)
Acronym: PREDICCMI
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2013/26
Record Dates: First submitted 2015-11-20; First posted 2015-12-22 (Estimated); Last update posted 2022-03-14 (Actual); Status verified 2022-03

CONDITIONS: Lower Limb Ischaemia
Keywords: Critical limb ischaemia; Peripheral occlusive arterial disease; Clinical prediction; Ankle pressure; Transcutaneous oxygen pressure; Toe pressure; Microcirculation
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia; Peripheral Arterial Occlusive Disease 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ICCMI: Patient hospitalized for lower limb arterial disease and suspected to have critical ischaemia
  Interventions: Other: Collection of clinical signs and symptoms

INTERVENTIONS:
Other: Collection of clinical signs and symptoms — Collection of clinical signs and symptoms used for developing a Clinical prediction rule of critical lower limb ischaemia (diagnosed by haemodynamic methods: ankle pressure, toe pressure-laser Doppler or photo-plethysmography, transcutaneous oxygen pressure) in patients with peripheral occlusive arterial disease

SUMMARY:
Critical limb ischaemia (CLI) is the most serious stage of peripheral occlusive arterial disease (POAD). Despite progress in the revascularization procedures, half these patients experience amputation or death after one year. One issue is to identify these subjects because aggressive treatment is necessary in those cases, while in others (ie leg ulcer in a patient with POAD but no rest lower limb ischaemia), revascularization will not be necessary. Then it would be useful to develop a simple score to help the physician to improve diagnosis of CLI.

DETAILED DESCRIPTION:
Today many patients with suspected critical limb ischaemia do not have objective assessment of limb ischaemia despite recommendations, mainly because of lack of vascular medicine units able to measure ischaemia with adequate methods such as toe pressure or TCpo2. It would be very useful to better identify the patients who need to be explored, or at least to have an evidence-based clinical assessment in those who cannot be explored . The objective is to develop a simple clinical prediction rule of critical lower limb ischaemia.

Two definitions are currently used for critical limb ischaemia. In both definitions, objective confirmation is needed for critical limb ischaemia by measurement of ankle pressure, toe pressure or transcutaneous oxygen pressure. These two latter measurements are mandatory in the numerous patients whose ankle pressure measurement is not possible (diabetes, chronic renal failure). Unfortunately few vascular medicine units exist to carry out these measurements, so that it would be useful to better identify those patients who need to be explored. In those who cannot be explored, better clinical assessment would also be very useful.

The investigators aim to develop a simple clinical prediction rule by completing a specific clinical chart in the patients hospitalized for peripheral occlusive arterial disease in Bordeaux, Toulouse and Limoges university hospital vascular medicine units and included in the COPART II cohort. Internal validation will be performed using cross-validation and bootstrap methods.

To achieve the secondary objective, the patients will be followed-up for the duration of the study (ie from 1 to 3 years) to evaluate the prediction of clinical outcomes (death or amputation) by both definitions of critical limb ischaemia.

ELIGIBILITY:
Inclusion Criteria:

* Patient coming for consultation or hospitalized for lower limb arterial disease and suspected to have critical ischaemia (ie rest pain or ulcer)

Non inclusion Criteria:

* Patient coming for consultation or hospitalized for lower limb arterial disease without rest pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized for peripheral occlusive arterial disease
Sampling Method: Non-Probability Sample
Enrollment: 603 (Actual)
Dates: Start 2016-02-15 (Actual); Primary Completion 2021-02-04 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Possible predictors: Clinical signs and symptoms collected on a specific clinical chart developed by investigators | Baseline (pre-inclusion visit)
  The specific clinical chart will be completed by 2 investigators independently in order to assess the reproductibility as well.
Predicted event: number of participants with diagnosis of Critical Lower Limb Ischaemia according to TASC I and II definitions | Day 1 (inclusion visit)

SECONDARY OUTCOMES:
Possible predictor: number of participants with diagnosis of Critical Lower Limb Ischaemia according to TASC I and II definitions | Day 1 (inclusion visit)
Predicted event: number of dead participants | Every year during study (up to 3 years)
  The vital status will be collected for every participant every year
Predicted event: number of participants who underwent amputation | Every year during study (up to 3 years)
  The amputation occurrence will be collected for every participant every year

CONTACTS AND LOCATIONS:
Overall Officials: Paul PEREZ, Study Chair — USMR, CHU de Bordeaux
Locations (3):
- France (3):
  - CHU de Bordeaux, Bordeaux
  - CHU de Limoges, Limoges
  - CHU de Toulouse, Toulouse